CLINICAL TRIAL: NCT03220516
Title: A Prospective Randomized Study Comparing Single-use Digital Flexible Ureteroscope, Nondisposable Fiber Optic and Digital Ureteroscope in Treatment of Upper Urinary Stone Less Than 2 cm
Brief Title: Single-use Digital Flexible Ureteroscope vs Nondisposable Fiber Optic vs Digital Ureteroscope
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Guohua Zeng (Other)
Collaborators: Dr. Lufti KIRDAR Kartal Research and training Hospital, Instanbul, Turkey (Unknown); Siloam St.Trudpert Hospital (Unknown)
Responsible Party: Sponsor-Investigator, Guohua Zeng, Doctor and Proffesor, The First Affiliated Hospital of Guangzhou Medical University
Organization: The First Affiliated Hospital of Guangzhou Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Scopes compared
Record Dates: First submitted 2017-07-01; First posted 2017-07-18 (Actual); Last update posted 2017-07-18 (Actual); Status verified 2017-07

CONDITIONS: Urolithiasis
MeSH Terms: conditions — Urolithiasis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- single-use digital ureteroscope (Experimental): Participants under this arm will undergo retrograde intrarenal surgery (RIRS) procedure under the single use digital ureteroscope.
  Interventions: Procedure: single use digital ureteroscope
- reusable fiberoptic ureteroscopes (Experimental): Participants under this arm will undergo the RIRS procedure under the reusable fiberoptic ureteroscope
  Interventions: Procedure: reusable fiberoptic ureteroscope
- reusable digital flexible ureteroscopes (Experimental): Participants under this arm will undergo the RIRS procedure under the reusable digital flexible ureteroscope.
  Interventions: Procedure: reusable digital flexible ureteroscope

INTERVENTIONS:
Procedure: single use digital ureteroscope — All participants in this arm will undergo RIRS using a single use digital ureteroscope.
  Arms: single-use digital ureteroscope
Procedure: reusable fiberoptic ureteroscope — All participants under this arm will undergo RIRS using a reusable fiberoptic ureteroscope
  Arms: reusable fiberoptic ureteroscopes
Procedure: reusable digital flexible ureteroscope — All participants under this arm will undergo RIRS using reusable digital flexible ureteroscope
  Arms: reusable digital flexible ureteroscopes

SUMMARY:
The aim of this trial is to compare the safety, efficacy and cost effectiveness of the three types of scopes.

DETAILED DESCRIPTION:
With the advancement of technology, flexible ureteroscopy (f-URS) has become an attractive option for surgical management of kidney stones. However, the durability of flexible ureteroscope still remains a major concern. Due to the high cost and limited durability, the cost-benefit of non-disposable flexible ureteroscope continues to be the most important factor for initiating and maintaining fURS programs worldwide, especially in the developing countries. Nowadays, disposable digital flexible ureteroscopes are available, offering an improved image resolution, no need for sterilization and repair, and more economic.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-70 years
2. American society of Anesthesiology (ASA) score 1 and 2
3. Renal or upper ureteral stone of diameter ≤ 2.0 cm

Exclusion Criteria:

1. Ureteral stricture, renal or ureteral deformity
2. Pregnancy
3. Patients with chronic kidney disease, CKD (serum creatine> 177 umol/L)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2017-08 (Estimated); Primary Completion 2020-09 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
cost of surgery | intraoperative
  the total cost of the procedure

SECONDARY OUTCOMES:
Stone free rate | 1month after surgery
stone free rate | 3months after surgery
complication rates | upto 3months
operative time | intraoperative
operator's satisfaction with the scope | intraoperative
  on the scope or 1-10